CLINICAL TRIAL: NCT07079579
Title: A Prospective, Single-arm, Open-label Study to Evaluate Different Initial Doses of Enarodustat Tablets for the Treatment of Anemia in Patients With Non-dialysis Chronic Kidney Disease
Brief Title: Enarodustat Tablets at Different Initial Doses for Anemia in Non-dialysis CKD Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAL0951A401
Record Dates: First submitted 2025-07-06; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Renal Anemia in Non-dialysis Chronic Kidney Disease
Keywords: Renal Anemia in Non-dialysis Chronic Kidney Disease; Enarodustat
MeSH Terms: interventions — enarodustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 2mg Enarodustat ESA-naïve (Experimental): ESA-naïve population initial phase：2mg QD for 4 weeks subsequent phase：1mg、2mg、4mg、6mg、8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Interventions: Drug: Enarodustat 2mg
- 3mg Enarodustat ESA-naïve (Experimental): ESA-naïve population initial phase：3mg QD for 4 weeks subsequent phase：1mg、2mg、4mg、6mg、8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Interventions: Drug: Enarodustat 3mg
- 4mg Enarodustat ESA-naïve (Experimental): ESA-naïve population initial phase：4mg QD for 4 weeks subsequent phase：1mg、2mg、4mg、6mg、8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Interventions: Drug: Enarodustat 4mg
- 2mg Enarodustat ESA-treated (Experimental): ESA-treated population initial phase：2mg QD for 4 weeks subsequent phase：1mg、2mg、4mg、6mg、8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Interventions: Drug: Enarodustat 2mg
- 3mg Enarodustat ESA-treated (Experimental): ESA-treated population initial phase：3mg QD for 4 weeks subsequent phase：1mg、2mg、4mg、6mg、8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Interventions: Drug: Enarodustat 3mg
- 4mg Enarodustat ESA-treated (Experimental): ESA-treated population initial phase：4mg QD for 4 weeks subsequent phase：1mg、2mg、4mg、6mg、8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Interventions: Drug: Enarodustat 4mg

INTERVENTIONS:
Drug: Enarodustat 2mg — initial phase：2mg QD for 4 weeks subsequent phase：1mg、2mg、4mg、6mg、8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Arms: 2mg Enarodustat ESA-naïve; 2mg Enarodustat ESA-treated
Drug: Enarodustat 3mg — initial phase：3mg QD for 4 weeks subsequent phase：1mg、2mg、4mg、6mg、8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Arms: 3mg Enarodustat ESA-naïve; 3mg Enarodustat ESA-treated
Drug: Enarodustat 4mg — initial phase：4mg QD for 4 weeks subsequent phase：1mg、2mg、4mg、6mg、8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Arms: 4mg Enarodustat ESA-naïve; 4mg Enarodustat ESA-treated

SUMMARY:
To evaluate the rationality of different initial doses of enarodustat for the treatment of anemia in ND-CKD patients

DETAILED DESCRIPTION:
The eligible subjects screened will be stratified by treatment history and randomized to the 2, 3, 4 mg dose groups in a 1:1:1 ratio. After receiving the initial doses of 2, 3, 4 mg/day for 4 weeks, the subjects will enter a 12-week maintenance treatment period with a total of 7 scheduled visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all the following criteria can be enrolled in this study:

  1. Male or female patients aged 18-75 years (inclusive);
  2. Body weight: 45-100 kg (inclusive);
  3. Stage 3-5 non-dialysis CKD complicated with renal anemia during the screening period, with an eGFR of 10-60 mL/min/1.73 m2 (exclusive) (calculated by CKD-EPI equation);
  4. Criteria for Hb levels at screening and baseline

  <!-- -->

  1. ESA-naïve population: Patients who do not receive ESA treatment in the past 12 weeks, with the Hb level greater than or equal to 70 g/L and less than 100 g/L;
  2. ESA-treated population: Patients who have received ESA treatment for at least 8 weeks, with the Hb level greater than or equal to 100 g/L and less than or equal to 120 g/L; 5.Female patients shall take contraceptive measures during the study; Patients who voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

* Patients who meet any one of the following criteria shall be excluded from the study:

  1. Patients with SF ≤100 μg/L and TSAT ≤20% at screening;
  2. Patients who are expected to start renal replacement therapy in the next 6 months as judged by the investigator;
  3. Patients with systemic hematologic disorders (e.g., myelodysplastic syndrome and aplastic anemia, etc.) or non-CKD-related anemia (hemolytic anemia, hemorrhagic anemia, cancer related anemia, etc.);
  4. Patients with a 1.5-fold increase in serum creatinine during the screening period;
  5. Patients who have received hypoxia-inducible factor prolyl hydroxylase inhibitors (HIF-PHI) within 8 weeks before screening;
  6. Patients with polycystic kidney disease;
  7. Patients with poorly controlled hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg at the screening visit);
  8. Patients with congestive cardiac failure (New York Heart Association [NYHA] Class III or above) or unstable angina;
  9. Patients who have experienced myocardial infarction, transient ischemic attack, cerebral infarction (except asymptomatic cerebral infarction) or venous thromboembolism (pulmonary embolism or deep vein thrombosis) from 24 weeks before screening to the first dose of the investigational drug;
  10. Patients with severe hepatobiliary disorders (e.g., AST or ALT >2.5 × upper limit of normal (ULN) at the screening visit, patients with hepatic cirrhosis or total bilirubin ≥1.5 × ULN at the screening visit);
  11. Patients who have received red blood cell transfusion from 12 weeks before screening to the first dose of the investigational drug;
  12. Patients who have received growth hormone, thyroid hormone, testosterone enanthate or methandienone from 12 weeks before screening to the first dose of the investigational drug;
  13. Patients who will undergo elective ophthalmic surgery in the next 6 months;
  14. Patients with severe hyperparathyroidism (e.g., iPTH ≥500 pg/mL at the screening visit);
  15. Patients with severe infections (e.g., active pulmonary tuberculosis and fungal infection, etc.);
  16. Patients suspected of having other non-infectious chronic inflammatory diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis and coeliac disease, etc.);
  17. Patients with a positive result for HIV, HCV or Treponema pallidum antibody, or with a positive result for HBsAg and HBV DNA ≥1,000 U/mL;
  18. Patients with a history of malignant tumors (including hematological malignancies) in the past 5 years;
  19. Patients with a history of severe drug allergy (e.g., anaphylactic shock) or hypersensitivity to other HIF-PHIs;
  20. Patients with a history of drug or alcohol abuse in the past two years;
  21. Patients who have received other investigational drugs (or study drugs) or received investigational medical devices (or study devices) from 12 weeks before the screening visit to the first dose of the investigational drug, or are participating in other interventional clinical studies (medical behaviors beyond routine diagnosis and treatment, implemented for study purposes) and receiving treatment;
  22. Patients who are pregnant, lactating or have the possibility of pregnancy (based on the results of the pregnancy test at the screening visit, the investigator cannot rule out the possibility of pregnancy);
  23. Patients with any medical conditions that, in the investigator's judgment, may pose a safety risk, may confound efficacy or safety evaluation, or may interfere with their participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean Hb level at Week 16 of treatment | week 16

SECONDARY OUTCOMES:
Cumulative proportion of subjects with Hb levels of ≥100 g/L and ≤120 g/L at each visit | week 0,2,4,8,12,16
Cumulative proportion of subjects with Hb levels of ≥110 g/L and <130 g/L at each visit | week 0,2,4,8,12,16
ESA-treated group: cumulative proportion of subjects with Hb levels ±10 g/L from baseline at Weeks 12-16 of treatment; | week12- 16
Hb levels at each visit | week 0,2,4,8,12,16
Change in Hb level from baseline at each visit | week 0,2,4,8,12,16
Dosage of administration of the investigational drug throughout the treatment period | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No